CLINICAL TRIAL: NCT05443698
Title: Sonograms Enable Looking Forward- Get Your iNformation 1 Trial
Brief Title: SELF-GYN1 (Sonograms Enable Looking Forward- Get Your iNformation 1 Trial)
Acronym: SELF-GYN1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turtle Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 016
Record Dates: First submitted 2022-06-22; First posted 2022-07-05 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Fertility Risk

STUDY DESIGN:
Intervention Model Description: Prospective, interventional, single arm clinical trial
Masking Description: Independent Readers reviewing Imaging Exams will be fully blinded to participant health history and exam setting.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Ultrasound Device (Other): All women who choose to enroll in the trial will undergo an at home transvaginal ultrasound guided by real-time remote supervision from a qualified and specially trained ultrasound technologist.
  Interventions: Device: Transvaginal ultrasound

INTERVENTIONS:
Device: Transvaginal ultrasound — Adult women in the U.S. who are eligible for the ultrasound trial on the basis of the inclusion/exclusion criteria will complete an at home transvaginal ultrasound guided by real-time remote supervision from a qualified and specially trained ultrasound technologist.

SUMMARY:
This clinical trial will evaluate the efficacy and safety of the use of the Turtle Health Ultrasound Scanner for the acquisition of transvaginal ultrasound images by a study participant, with no previous training, in her home when guided by real-time remote supervision from a qualified and specially trained ultrasound technologist.

DETAILED DESCRIPTION:
Those images will be assessed for their image quality by qualified Independent Readers. The study is intended to assess the ability of at home imaging performed with the Turtle Health Ultrasound Scanner to reliably produce quality images as compared to objective performance criteria set by the American Institute of Ultrasound in Medicine (AIUM).

The clinical investigation is intended to extend the findings of a published trial (SELF-HELP) to real-world performance.

Each participant will have imaging performed at-home. The at-home imaging will be conducted using the Turtle Health Ultrasound Scanner, manipulated by the participant and guided in real time by a remote ultrasound technologist that has received special training with the device. Home imaging will follow the procedures included in planned device labeling. Imaging obtained will include, at minimum, each of the specific imaging views and components defined in the "American Institute of Ultrasound in Medicine (AIUM) Case Study Submission Requirements: Gynecologic Ultrasound".

Imaging Scans will be assessed by at least two (2) independent readers who are physicians expert in the interpretation of transvaginal ultrasound gynecologic imaging studies. Images will have participant name redacted and each independent reader will be blinded to any participant information other than the images themselves. They will also be blinded to the assessments of the other readers. In-clinic Imaging Scans obtained from either or both of previous trials and in-clinic scans will be included in rating batches for calibration.

ELIGIBILITY:
Inclusion Criteria:

* Woman, as defined by sex at birth
* Age 22 years or older at the time of eligibility screening
* Premenopausal
* BMI < 40 kg/m2
* Unlikely to be pregnant during home scan, based on either current intrauterine device (IUD) or other birth control use or recent menstruation, defined as the home scan occurring between day 3 and 10 of the menstrual cycle based on patient self-report
* English-speaking and able to follow verbal instructions of the remote ultrasound technologist as determined by the ability to complete the consent process unassisted
* Ability to manipulate a 1 lb. weight by hand
* Residence in state where a PI holds a valid license to practice medicine
* Ability to receive signature delivery of the investigational ultrasound device
* Ability to return the investigational ultrasound device by specified instructions

Exclusion Criteria:

* Pregnant or may be pregnant
* Has recently given birth, and has had fewer than 3 postpartum menstrual cycles
* Has recently had a stillbirth or abortion more than 20 weeks (subject to the 3 postpartum menstrual cycles above). Miscarriages or abortions less than 20 weeks are subject to two wait cycles
* Has changed birth control within the current menstrual cycle (one 'washout' cycle is required)
* Turtle Health employees
* Has known cancer of a pelvic organ, not currently in remission
* Not able to schedule a scan while meeting the requirements above prior to the end of the trial. For example, women who change birth control within the last cycle of the trial (and would require a 'washout cycle' that would delay trial close) or who are unable to schedule within the last few weeks of the trial after reasonable scheduling efforts have been made
* Previous hysterectomy or oophorectomy
* Does not have one or more of the following anatomic organs: vagina, left ovary, right ovary, or uterus
* Subjects with prior scanning experience are included in the trial (as they would be in the real world) but excluded from the primary image quality endpoint (due to experience potentially influencing that endpoint) and analyzed separately as a subgroup for that endpoint only. This sub-population is capped at 200 subjects (~20% of trial)

Min Age: 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Woman, as defined by sex at birth
Enrollment: 365 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
Image Quality | 6 weeks
  Each Independent Reader will make a determination of whether each Imaging Scan is of 'diagnostic quality' or 'not diagnostic quality', in its totality, for the purpose of a diagnostic gynecological ultrasound examination.
Net Promoter Score (NPS) | 6 weeks
  All subjects will be asked to complete the question 'How likely are you to recommend the experience to a friend or colleague?.' It is expected that a high share of patients will report a positive NPS.

SECONDARY OUTCOMES:
False Positives | 6 weeks
  Rate of false positives of 'significant findings'
Performance Task of Independent Readers | 6 weeks
  Each Independent Reader will assess the suitability of the Imaging Study for use on each of ten specific imaging tasks defined by the AIUM practice parameters as required for a high quality two-dimensional gynecological ultrasound imaging study.
Box Opening | 6 weeks
  Patient opens box at correct time (not early)
Patient Identifier | 6 weeks
  Correct patient is identified by tech and tests (not wrong patient)
Probe Cover | 6 weeks
  Patient correctly applies probe cover and uses it successfully during the scan
Correct Cavity | 6 weeks
  Patient places probe in correct cavity (vaginal vs. anal)
Timely Return | 6 weeks
  Patient ships product back in a timely fashion
Shipping Damage | 6 weeks
  Rate at which probe is damaged in transit
Successful Return | 6 weeks
  Rate at which probe remains in working condition and able to be reprocessed
Minor Pain or Discomfort | 6 weeks
  Rate at which subjects report minor pain, discomfort, or similarly mild symptoms lasting under 24 hours
All Other Adverse Events | 6 weeks
  Rate at which subjects report adverse events, side effects, or other sequelae other than minor pain, discomfort, or similarly mild symptoms lasting under 24 hours
Successful Reprocessing | 6 weeks
  Number of probes undergoing reprocessing that are reprocessed properly per internal standard operating procedures
Ultrasound technologist satisfaction | 6 months
  Difference in average weekly satisfaction between in-person and virtual settings based on survey responses
Ultrasound technologist availability | 6 months
  Estimation of weekly increase in personnel capacity enabled by device based on number of ultrasound technologists available.
Ultrasound technologist safety | 6 months
  Implied/potential estimation of injury reduction based on survey results
Correct setting of care guess rate | 6 months
  Including in-clinic 'control' data from previous study or from in-clinic scans with same device
Sub-group exploratory endpoints: Endpoint 1 | 1 year
  Results from the primary end point "Image Quality" will also be reported by sub-populations of interest. The sub-populations are:
  1. Class I obese patients (BMI between 30 and 35, inclusive)
  2. Class II+ obese patients (BMI greater than 35)
  3. Aged 40 or older
  4. Residing in 'completely rural' or 'mostly rural' counties
  5. Symptoms indicating possible pathology (where available)
  6. No record of visiting a doctor in the 24 months prior to enrollment (where available)
  7. Educational attainment less than some college
  8. Identifying as Hispanic or Latino
  9. Identifying as
     * American Indian or Alaska Native
     * Asian
     * Black or African American
     * Native Hawaiian or Other Pacific Islander
     * White
     * Multiple identities selected
Sub-group exploratory endpoints: Endpoint 2 | 1 year
  Results from the primary end point "Net Promoter Score (NPS)" will also be reported by sub-populations of interest. There sub-populations are:
  1. Class I obese patients (BMI between 30 and 35, inclusive)
  2. Class II+ obese patients (BMI greater than 35)
  3. Aged 40 or older
  4. Residing in 'completely rural' or 'mostly rural' counties
  5. Symptoms indicating possible pathology (where available)
  6. No record of visiting a doctor in the 24 months prior to enrollment (where available)
  7. Educational attainment less than some college
  8. Identifying as Hispanic or Latino
  9. Identifying as
     * American Indian or Alaska Native
     * Asian
     * Black or African American
     * Native Hawaiian or Other Pacific Islander
     * White
     * Multiple identities selected

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Virtual Site, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chung EH, Petishnok LC, Conyers JM, Schimer DA, Vitek WS, Harris AL, Brown MA, Jolin JA, Karmon A, Styer AK. Virtual Compared With In-Clinic Transvaginal Ultrasonography for Ovarian Reserve Assessment. Obstet Gynecol. 2022 Apr 1;139(4):561-570. doi: 10.1097/AOG.0000000000004698. Epub 2022 Mar 10. PMID 35271530
- [Background] Birch Petersen K, Maltesen T, Forman JL, Sylvest R, Pinborg A, Larsen EC, Macklon KT, Nielsen HS, Hvidman HW, Nyboe Andersen A. The Fertility Assessment and Counseling Clinic - does the concept work? A prospective 2-year follow-up study of 519 women. Acta Obstet Gynecol Scand. 2017 Mar;96(3):313-325. doi: 10.1111/aogs.13081. Epub 2017 Feb 3. PMID 27990627
- [Background] Farquhar C, Ekeroma A, Furness S, Arroll B. A systematic review of transvaginal ultrasonography, sonohysterography and hysteroscopy for the investigation of abnormal uterine bleeding in premenopausal women. Acta Obstet Gynecol Scand. 2003 Jun;82(6):493-504. doi: 10.1034/j.1600-0412.2003.00191.x. PMID 12780419